CLINICAL TRIAL: NCT04771273
Title: Multicenter, Double-blind, Parallel-group, Randomized, 48 Weeks, Dose-ranging, Placebo-controlled Phase II Trial to Evaluate Efficacy, Safety and Tolerability of Multiple Subcutaneous (s.c.) Doses of BI 456906 in Patients With Non-alcoholic Steatohepatitis (NASH) and Fibrosis.
Brief Title: A Study to Test Safety and Efficacy of Survodutide (BI456906) in Adults With Non-alcoholic Steatohepatitis (NASH) and Fibrosis (F1-F3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0043; 2020-002723-11 (EudraCT Number)
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Survodutide 2.4 mg - planned maintenance treatment (Experimental)
  Interventions: Drug: Survodutide
- Survodutide 4.8 mg - planned maintenance treatment (Experimental)
  Interventions: Drug: Survodutide
- Survodutide 6.0 mg - planned maintenance treatment (Experimental)
  Interventions: Drug: Survodutide
- Placebo - planned maintenance treatment (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Survodutide — Survodutide
  Other Names: BI 456906
  Arms: Survodutide 2.4 mg - planned maintenance treatment; Survodutide 4.8 mg - planned maintenance treatment; Survodutide 6.0 mg - planned maintenance treatment
Drug: Placebo — Placebo
  Arms: Placebo - planned maintenance treatment

SUMMARY:
This study is open for men and women with a liver disease called nonalcoholic steatohepatitis (NASH) and liver fibrosis. The purpose of the study is to find out whether a medicine called BI 456906 helps patients with NASH and liver fibrosis. The study tests 3 different doses of BI 456906 to find the dose that helps best. Participants are put into 4 groups randomly, which means by chance. There are 3 groups that each receive a different dose of BI 456906 and there is 1 group that receives placebo. BI 456906 and placebo are given as an injection under the skin once per week. The placebo injection looks like the BI 456906 injection but does not contain any medicine.

Participants are in the study for a little over 1 year (60 weeks). During this time, they visit the study site several times and have some video calls in addition. At the visits, the study doctors take different measurements. To see whether the treatment works, the doctors take a very small sample of liver tissue (biopsy) from each participant at the start and at the end of the study. They also examine the liver by ultrasound and MRI. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years (or who are of legal age in countries where that is greater than 18 years) and ≤ 80 years of age at time of consent.
2. Diagnosis of non-alcoholic steatohepatitis (NASH) (Non-alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) ≥ 4, with at least 1 point in inflammation and ballooning each) and fibrosis stage F1-F3 proven by a biopsy conducted during the screening period or by a historical biopsy conducted within the last 6 months prior to randomization and stable body weight defined as less than 5% self-reported change in body weight between the historical biopsy and randomization, if a historical biopsy is used.
3. Liver fat fraction ≥ 8% measured by Magnetic Resonance Imaging (MRI)-Proton Density Fat Fraction (PDFF) and liver stiffness > 6.0 kPa measured by FibroScan® at Visit 1 (if biopsy is scheduled during the screening period MRI-PDFF and FibroScan® assessments have to be performed prior to the biopsy). However, the diagnosis of NASH and fibrosis at liver biopsy (including historical biopsy) is the primary assessment to establish patient eligibility.
4. Patients willing and able to undergo liver biopsies per protocol as judged by the Investigator.
5. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
6. Women of childbearing potential (WOCBP)1 must be willing and able to use two forms of effective contraception where at least one form is highly effective methods of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

Further inclusion criteria apply.

Exclusion Criteria:

1. Current or history of significant alcohol consumption (defined as intake of > 210 g/ week in males and > 140 g/ week in females on average over a consecutive period of more than 3 months) or inability to reliably quantify alcohol consumption based on Investigator judgement within the last 5 years.
2. Intake of medications historically associated with liver injury, hepatic steatosis or steatohepatitis within 12 weeks prior to Visit 1. Intake of restricted medications or any medications considered likely to interfere with the safe conduct of the trial.
3. History of other forms of chronic liver disease (e.g., viral hepatitis, autoimmune liver disease, primary biliary sclerosis, primary sclerosing cholangitis, Wilson's disease, hemochromatosis, Alpha-1 Antitrypsin (A1At) deficiency, history of liver transplantation). Hepatitis B and C testing will be done at Visit 1. Patients with positive Hepatitis B surface antigen (HBsAg) should be excluded. Patients treated for hepatitis C must have a negative RNA test at screening and also be Hepatitis C Virus (HCV) RNA negative for at least 3 years prior to screening in order to be eligible for the trial.
4. Suspicion, diagnosis, or history of hepatocellular carcinoma (HCC), or any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
5. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, manifest hypo- or hyperthyroidism at Visit 1.
6. History of chronic or acute pancreatitis or elevation of serum lipase/amylase > 2x ULN or fasting serum triglyceride levels of > 500 mg/dL (> 5.65 mmol/L) at screening.
7. Known history of HIV (Human Immunodeficiency Virus) infection and/or tuberculosis and/or an acute COVID-19 infection at Visit 1 (confirmed by SARS CoV-2 RT-PCR test). Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (154):
- United States (36):
  - North Alabama Health Research, LLC, Huntsville, Alabama
  - Southern California Research Center, Coronado, California
  - Velocity Clinical Research, Huntington Park, California
  - Velocity Clinical Research, Panorama City, California
  - Quest Clinical Research, San Francisco, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Integrity Clinical Research, LLC, Doral, Florida
  - Covenant Metabolic Specialists, LLC, Fort Myers, Florida
  - Optimus U Corporation, Miami, Florida
  - Sanchez Clinical Research ,Inc, Miami, Florida
  - Ocala GI Research, Ocala, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - National Diabetes and Obesity Research Institute, Biloxi, Mississippi
  - Gastrointestinal Associates, Flowood, Mississippi
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - Northeast GI Research Division, Concord, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Digestive Diseases Research Center, Greenwood, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Digestive Health Research, LLC, Hermitage, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Texas Liver Institute, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Houston Methodist Hospital, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Gold Coast University Hospital, Southport, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (3):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
- Edegem - UNIV UZ Antwerpen, Edegem, Belgium
- Canada (3):
  - University Hospital (LHSC), London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
- China (13):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - NanFang Hosptial, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - First People's hospital of Yunann Province, Kunming
  - The Second Hospital of Nanjing, Nanjing
  - Shanghai Public Health Clinical Center, Shanghai
  - Tianjin Third Central Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Med College, Wenxzhou
- Czechia (2):
  - Regional Hospital Liberec, Liberec
  - General Faculty Hospital, Prague, Prague
- France (4):
  - HOP l'Archet, Nice
  - HOP La Pitié Salpêtrière, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Civil, Strasbourg
- Germany (9):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Synexus Clinical Research GmbH, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Synexus Clinical Research GmbH, Frankfurt
  - Synexus Clinical Research GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - Attikon University Hospital, Haidari-Athens
  - General Hospital of Thessaloniki "Hippokrateio", Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (3):
  - Synexus Hungary Healthcare Service Ltd., Budapest
  - Fed.St. Istvan&Szent Laszlo Hospital, Budapest
  - Synexus Hungary Healthcare Service Ltd, Gyula
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Western Galilee Hospital, Nahariya
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (6):
  - Ospedale Civile di Baggiovara, Baggiovara (MO)
  - A.O. Univ. Policlinico "Paolo Giaccone", Palermo
  - Poli Univ A. Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - IRCCS Ospedale "Casa Sollievo della Sofferenza", SAN Giovanni Rotondo (FG)
  - AO Città della Salute e Scienza, Torino
- Japan (21):
  - Ehime University Hospital, Ehime, Toon
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - Kurume University Hospital, Fukuoka, Kurume
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - National Hospital Organization Yokohama Medical Center, Kanagawa, Yokohama
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Shinshu University Hospital, Nagano, Matsumoto
  - Nagano Municipal Hospital, Nagano, Nagano
  - Nara Medical University Hospital, Nara, Kashihara
  - Suita Hospital, Osaka, Suita
  - Saga University Hospital, Saga, Saga
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Juntendo University Shizuoka Hospital, Shizuoka, Izunokuni
  - Tokyo Medical and Dental University Hospital, Tokyo, Bunkyo-ku
- Malaysia (3):
  - Universiti Sains Malaysia Hospital, Kelantan
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
- Netherlands (3):
  - Amsterdam UMC, location VUMC, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Sint Franciscus, Locatie Vlietland, Rotterdam
- New Zealand (2):
  - New Zealand Clinical Research (NZCR), Auckland
  - Middlemore Clinical Trials, Papatoetoe
- Poland (11):
  - INTERCORE Medical Center, Bydgoszcz
  - Synexus Poland, Branch in Czestochowa, Częstochowa
  - Private health care facility "Your Health EL" LLC, Elblag
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Gdynia
  - University Clinical Center Professor Gibinskiego, Katowice
  - University Hospital in Krakow, Krakow
  - Medicome Limited Liability Company, Oświęcim
  - Centrum Medyczne Synexus, Warsaw
  - Synexus Poland, Branch in Wroclaw, Wroclaw
  - ETG Zamosc, Zamość
- Portugal (2):
  - ULS de Santa Maria, E.P.E, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (3):
  - Pusan National Univ. Hosp, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Hospital, Seoul
- Spain (6):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital de Montecelo, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
- Taiwan (4):
  - Chia Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Chen Kung University, Dept of Neurology, Tainan
  - Chang Gung Memorial Hospital(Linkou), Taoyuan
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Synexus - Hexham, Hexham
  - Aintree University Hospital, Liverpool
  - King's College Hospital, London
  - Queen's Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Sanyal AJ, Bedossa P, Fraessdorf M, Neff GW, Lawitz E, Bugianesi E, Anstee QM, Hussain SA, Newsome PN, Ratziu V, Hosseini-Tabatabaei A, Schattenberg JM, Noureddin M, Alkhouri N, Younes R; 1404-0043 Trial Investigators. A Phase 2 Randomized Trial of Survodutide in MASH and Fibrosis. N Engl J Med. 2024 Jul 25;391(4):311-319. doi: 10.1056/NEJMoa2401755. Epub 2024 Jun 7. PMID 38847460
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 48 weeks, multi-centre, randomised, dose-ranging, double-blind, placebo-controlled, parallel-group trial to evaluate efficacy, safety and tolerability of multiple subcutaneous (s.c.) doses of survodutide (BI 456906) in patients with non-alcoholic steatohepatitis (NASH).
  Main parameters for inclusion of patients and for evaluation of treatment response were based on the histological evaluation from the liver biopsy and non-invasive imaging modalities.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Patients who met the eligibility criteria at an initial screening visit had a second screening visit for biopsy to confirm their eligibility, if no sufficient material from a historical biopsy within the 6 months prior to randomisation was available.
Groups:
- Survodutide 2.4 mg - Planned Maintenance Treatment: Patients with non-alcoholic steatohepatitis (NASH) with non-alcoholic fatty liver disease (NAFLD) activity score (NAS) ≥4 and fibrosis stage 1-3 (F1-F3). were to be administered once weekly, subcutaneously a solution for injection of survodutide at a starting dose of 0.3 milligrams (mg) followed by a dose escalation up to the maintenance dose of 2.4 mg of survodutide.
  The total treatment duration was 48 weeks (consisting of up to 24 weeks dose escalation period and at least 24 weeks maintenance period).
  Participants not tolerating the assigned dose due to gastrointestinal adverse events had the option of a dose adjustment which could lead to a maintenance dose lower than the dose the patient was randomized to.
- Survodutide 4.8 mg - Planned Maintenance Treatment: Patients with non-alcoholic steatohepatitis (NASH) with non-alcoholic fatty liver disease (NAFLD) activity score (NAS) ≥4 and fibrosis stage 1-3 (F1-F3). were to be administered once weekly, subcutaneously a solution for injection of survodutide at a starting dose of 0.3 milligrams (mg) followed by a dose escalation up to the maintenance dose of 4.8 mg of survodutide.
  The total treatment duration was 48 weeks (consisting of up to 24 weeks dose escalation period and at least 24 weeks maintenance period).
  Participants not tolerating the assigned dose due to gastrointestinal adverse events had the option of a dose adjustment which could lead to a maintenance dose lower than the dose the patient was randomized to.
- Survodutide 6.0 mg - Planned Maintenance Treatment: Patients with non-alcoholic steatohepatitis (NASH) with non-alcoholic fatty liver disease (NAFLD) activity score (NAS) ≥4 and fibrosis stage 1-3 (F1-F3). were to be administered once weekly, subcutaneously a solution for injection of survodutide at a starting dose of 0.3 milligrams (mg) followed by a dose escalation up to the maintenance dose of 6.0 mg of survodutide.
  The total treatment duration was 48 weeks (consisting of up to 24 weeks dose escalation period and at least 24 weeks maintenance period).
  Participants not tolerating the assigned dose due to gastrointestinal adverse events had the option of a dose adjustment which could lead to a maintenance dose lower than the dose the patient was randomized to.
- Placebo - Planned Maintenance Treatment: Patients with non-alcoholic steatohepatitis (NASH) with non-alcoholic fatty liver disease (NAFLD) activity score (NAS) ≥4 and fibrosis stage 1-3 (F1-F3). were administered once weekly, subcutaneously a solution for injection of placebo matching survodutide. The total treatment duration was 48 weeks (consisting of up to 24 weeks dose escalation period and at least 24 weeks maintenance period).
Period: Dose Escalation Period
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Started (Randomised) | 73 | 73 | 75 | 74
Treated With Trial Medication | 73 | 72 | 74 | 74
Completed (Completed treatment with trial medication) | 62 | 63 | 57 | 68
Not Completed | 11 | 10 | 18 | 6
Not completed — Not treated with trial medication | 0 | 1 | 1 | 0
Not completed — Other reasons than listed | 2 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 3 | 1
Not completed — Burden of study procedures | 1 | 0 | 0 | 0
Not completed — Change of residence | 0 | 0 | 0 | 1
Not completed — Perceived lack of efficacy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 8 | 9 | 12 | 2
Period: Maintenance Period
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Started | 62 | 63 | 57 | 68
Completed (Completed treatment with trial medication) | 53 | 55 | 49 | 64
Not Completed | 9 | 8 | 8 | 4
Not completed — Other than listed | 4 | 2 | 0 | 3
Not completed — Burden of study procedures | 1 | 0 | 0 | 0
Not completed — Change of residence | 0 | 1 | 3 | 0
Not completed — Perceived lack of efficacy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 5 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Treated set - planned maintenance treatment: included all patients that were administered survodutide or placebo matching survodutide. Patients are analyzed according to the planned treatment (planned maintenance dose strength) they were assigned at randomisation even if patients did not reach the maintenance period at all, and therefore did not "settle" on any maintenance dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment | Total
Number analyzed (Participants) | 73 | 72 | 74 | 74 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (13.7) | 50.2 (12.9) | 50.4 (13.1) | 53.0 (11.5) | 50.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 41 | 44 | 155
  Male | 37 | 38 | 33 | 30 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 19 | 26 | 22 | 81
  Not Hispanic or Latino | 59 | 53 | 48 | 52 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 24 | 22 | 17 | 17 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 2 | 3 | 0 | 0 | 5
  White | 46 | 47 | 56 | 56 | 205
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
NAS score at baseline [Mean (Standard Deviation); unit: score on a scale] — The non-alcoholic fatty liver disease (NAFLD) activity score (NAS) represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
  score on a scale | 5.2 (1.0) | 5.3 (1.1) | 5.1 (1.0) | 5.2 (1.1) | 5.2 (1.0)
Number of participants at each category of liver fibrosis stage at baseline [Count of Participants; unit: Participants] — Number of participants at each category of liver fibrosis stage at baseline is reported.
  The total score for the fibrosis stage ranges from 0 to 4 with higher score indication worsening of the disease and the stages of fibrosis based on their location are the following:
  * 1A Zone 3, perisinusoidal, delicate;
  * 1B Zone 3, perisinusoidal, dense;
  * 1C Portal, periportal only;
  * 2 Zone 3, perisinusoidal + portal, periportal only;
  * 3 Bridging fibrosis;
  * 4 Cirrhosis.
  Participants
    Stage 1A | 0 | 3 | 3 | 2 | 8
    Stage 1B | 17 | 7 | 14 | 9 | 47
    Stage 1C | 3 | 3 | 6 | 3 | 15
    Stage 2 | 30 | 36 | 24 | 30 | 120
    Stage 3 | 23 | 23 | 27 | 30 | 103
Number of participants in each category of diabetes at baseline [Count of Participants; unit: Participants] — Number of participants at each category of diabetes at baseline is reported. The reported categories of diabetes stratification are the following: Yes, No.
  Participants
    No | 44 | 43 | 44 | 45 | 176
    Yes | 29 | 29 | 30 | 29 | 117
Number of patients in each category of NAS score [Count of Participants; unit: Participants] — Number of patients in each category of non-alcoholic fatty liver disease (NAFLD) activity score (NAS) score is reported. The NAS represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease. The reported categories of NAS score range are: 0; 1; 2; 3; 4; 5; 6; 7; 8.
  Participants
    0 | 0 | 0 | 0 | 0 | 0
    1 | 0 | 0 | 0 | 0 | 0
    2 | 0 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0 | 0
    4 | 21 | 20 | 26 | 22 | 89
    5 | 27 | 21 | 17 | 28 | 93
    6 | 17 | 22 | 26 | 8 | 73
    7 | 8 | 8 | 5 | 16 | 37
    8 | 0 | 1 | 0 | 0 | 1
Number of patients in each category of the NAS sub-scores (steatosis and lobular inflammation) [Count of Participants; unit: Participants] — The non-alcoholic fatty liver disease (NAFLD) activity score (NAS) represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
  Number of patients in each category of the score range for steatosis and lobular inflammation is reported.
  Participants
    Steatosis: 0 | 0 | 0 | 0 | 0 | 0
    Steatosis: 1 | 6 | 0 | 1 | 3 | 10
    Steatosis: 2 | 38 | 38 | 49 | 43 | 168
    Steatosis: 3 | 29 | 34 | 24 | 28 | 115
    Lobular inflammation: 0 | 0 | 0 | 0 | 0 | 0
    Lobular inflammation: 1 | 32 | 31 | 36 | 37 | 136
    Lobular inflammation: 2 | 38 | 40 | 36 | 32 | 146
    Lobular inflammation: 3 | 3 | 1 | 2 | 5 | 11
Number of patients in each category of the NAS sub-scores (ballooning) [Count of Participants; unit: Participants] — The non-alcoholic fatty liver disease (NAFLD) activity score (NAS) represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
  Number of patients in each category of the score range for ballooning is reported.
  Participants
    0 | 0 | 0 | 0 | 0 | 0
    1 | 55 | 55 | 53 | 49 | 212
    2 | 18 | 17 | 21 | 25 | 81

OUTCOME MEASURES:

1. Primary Outcome: Improvement (Yes/ no) From Baseline in Liver Histological Findings Based on Liver Biopsy After 48 Weeks of Treatment in Patients With NASH (NAS ≥ 4, Fibrosis F1-F3) - Actual Maintenance Treatment
Description: Percentage of patients who had an improvement from baseline in liver histological findings based on liver biopsy after 48 weeks of treatment is reported. Percentages were rounded to one decimal place.
  Improvement in histological findings was defined as a composite of improvement in NASH and no worsening of fibrosis.
  Improvement in non-alcoholic steatohepatitis (NASH) was defined as decrease of at least 2 points in non-alcoholic fatty liver disease (NAFLD) activity score (NAS) with at least 1 point decrease in NAS subscore of either lobular inflammation or ballooning.
  The NAS represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
  The total score for the fibrosis stage ranges from 0 to 4 with higher score indication worsening of the disease.
  Patients without post-baseline data were considered non-responders.
Time Frame: At baseline and at 48 weeks.
Population: Treated set - actual maintenance treatment. Patients are analyzed according to the actual treatment they received at the start of the dose maintenance period (for patients who reached the maintenance period) or the next maintenance dose up from the dose at treatment discontinuation (for patients who discontinued treatment prior to the maintenance period).
Measure: Number; unit: Percentage of participants
Groups:
- Survodutide 2.4 mg - Actual Maintenance Treatment: This arm includes patients who were treated with 2.4 mg of survodutide administered weekly at the start of the maintenance period, for patients who reached the maintenance period, regardless of whether this was the randomised (planned) dose or not, and regardless of whether the patient stayed on that dose throughout the maintenance period.
  This arm includes also those patients for whom the next maintenance dose up from the dose at treatment discontinuation was 2.4 mg of survodutide administered weekly, for patients who discontinued treatment prior to the maintenance period, regardless of the reason for the treatment discontinuation.
- Survodutide 4.8 mg - Actual Maintenance Treatment: This arm includes patients who were treated with 4.8 mg of survodutide administered weekly at the start of the maintenance period, for patients who reached the maintenance period, regardless of whether this was the randomised (planned) dose or not, and regardless of whether the patient stayed on that dose throughout the maintenance period.
  This arm includes also those patients for whom the next maintenance dose up from the dose at treatment discontinuation was 4.8 mg of survodutide administered weekly, for patients who discontinued treatment prior to the maintenance period, regardless of the reason for the treatment discontinuation.
- Survodutide 6.0 mg - Actual Maintenance Treatment: This arm includes patients who were treated with 6.0 mg of survodutide administered weekly at the start of the maintenance period, for patients who reached the maintenance period, regardless of whether this was the randomised (planned) dose or not, and regardless of whether the patient stayed on that dose throughout the maintenance period.
  This arm includes also those patients for whom the next maintenance dose up from the dose at treatment discontinuation was 6.0 mg of survodutide administered weekly, for patients who discontinued treatment prior to the maintenance period, regardless of the reason for the treatment discontinuation.
- Placebo - Actual Maintenance Treatment: This arm includes patients who were treated with placebo matching survodutide administered weekly at the start of the maintenance period, for patients who reached the maintenance period, regardless of whether this was the randomised (planned) dose or not, and regardless of whether the patient stayed on that dose throughout the maintenance period.
  This arm includes also those patients who were receiving Placebo matching survodutide administered weekly and who discontinued treatment prior to the maintenance period, regardless of the reason for the treatment discontinuation.
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 93 | 69 | 52 | 79
Percentage of participants | 38.7 | 63.8 | 55.8 | 15.2
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; The logistic regression model included actual treatment, presence of diabetes of any type and Baseline Fibrosis Score. Firth's penalized regression was used; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0010, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 3.47, 95% CI 2-sided [1.66 to 7.25] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < 0.0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 9.52, 95% CI 2-sided [4.35 to 20.85] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 7.07, 95% CI 2-sided [3.10 to 16.16]
Statistical Analysis 4: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; A flat vs. non-flat dose-response relationship across the 3 doses of survodutide and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 6 different plausible dose-response patterns (linear, exponential1, exponential2, Emax1, Emax2, quadratic) while keeping full control of the type I error (one-sided alpha of 0.050); Test type: Other — Logistic regression estimates were used as input for the MCP-Mod. The logistic regression model was fitted without an intercept, and included presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3] and the dose group as factors. P-values from the contrast tests corresponding to each dose response pattern evaluated were adjusted for the multiple comparisons performed; p < 0.0001, MCP-Mod linear model fit; Linear model fit assumption
Statistical Analysis 5: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p < 0.0001, MCP-Mod exponential-1 model fit; Model assumption: 25% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 6: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — Logistic regression estimates were used as input for the MCP-Mod. The logistic regression model was fitted without an intercept and included presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3] and the dose group as factors. P-values from the contrast tests corresponding to each dose response pattern evaluated were adjusted for the multiple comparisons performed; p = 0.0008, MCP-Mod exponential -2 model fit; Model assumption: 5% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 7: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 6]; p < 0.0001, MCP-Mod Emax1 model fit; Model assumption: 50% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 8: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 6]; p < 0.0001, MCP-Mod Emax2 model fit; Model assumption: 80% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 9: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 6]; p < 0.0001, MCP-Mod quadratic model fit; Model assumption: Maximum effect is achieved at dose 4.8 mg

2. Primary Outcome: Improvement (Yes/ no) From Baseline in Liver Histological Findings Based on Liver Biopsy After 48 Weeks of Treatment in Patients With NASH (NAS ≥ 4, Fibrosis F1-F3) - Planned Maintenance Treatment
Description: Percentage of patients who had an improvement from baseline in liver histological findings based on liver biopsy after 48 weeks of treatment is reported. Percentages were rounded to one decimal place.
  Improvement in histological findings was defined as a composite of improvement in non-alcoholic steatohepatitis (NASH) and no worsening of fibrosis.
  Improvement in NASH was defined as decrease of at least 2 points in non-alcoholic fatty liver disease (NAFLD) activity score (NAS) with at least 1 point decrease in NAS subscore of either lobular inflammation or ballooning.
  The NAS represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
  The total score for the fibrosis stage ranges from 0 to 4 with higher score indication worsening of the disease.
  Patients without post-baseline data were considered non-responders.
Time Frame: At baseline and after 48 weeks of treatment.
Population: Treated set - planned maintenance treatment: included all patients that were administered survodutide or placebo matching survodutide. Patients are analyzed for this endpoint according to the planned treatment (planned maintenance dose strength) they were assigned at randomisation even if patients did not reach the maintenance period at all, and therefore did not "settle" on any maintenance dose.
Measure: Number; unit: percentage of participants
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 73 | 72 | 74 | 74
percentage of participants | 46.6 | 62.5 | 43.2 | 13.5
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; The logistic regression model includes planned treatment, presence of diabetes of any type and Baseline Fibrosis Score. Firth's penalized regression was used; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 5.49, 95% CI 2-sided [2.46 to 12.28] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 10.14, 95% CI 2-sided [4.49 to 22.87] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 4.87, 95% CI 2-sided [2.18 to 10.91] — Survodutide 6.0 mg vs. Placebo
Statistical Analysis 4: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 6]; p = 0.0001, MCPMod linear model fit; linear model fit assumption
Statistical Analysis 5: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.0115, MCPMod exponential-1 model fit; Model assumption: 25% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 6: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.2204, MCP-Mod exponential-2 model fit; Model assumption: 5% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 7: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p < 0.0001, MCP-Mod Emax1 model fit; Model assumption: 50% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 8: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 6]; p < 0.0001, MCP-Mod Emax2; Model assumption: 80% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 9: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p < 0.0001, MCP-Mod quadratic model fit; Model assumption: Maximum effect is achieved at dose 4.8 mg

3. Secondary Outcome: Improvement of Liver Fat Content (Yes/ no) Defined as at Least 30% Relative Reduction in Liver Fat Content After 48 Weeks of Treatment Compared to Baseline Assessed by MRI-PDFF - Actual Maintenance Treatment
Description: Percentage of participants with improvement in liver fat content is reported. Improvement in liver fat content was defined as percentage reduction from baseline of ≥30% in liver fat content after 48 weeks of treatment compared to baseline. Percentages were rounded to one decimal place.
  Liver fat content was assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF).
  Patients without post-baseline values were imputed as non-responders.
Time Frame: At baseline and after 48 weeks.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 93 | 69 | 52 | 79
Percentage of participants | 50.5 | 66.7 | 76.9 | 16.5
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; The logistic regression model included actual treatment, presence of diabetes of any type, baseline liver fat content and baseline fibrosis score. Firth's penalized regression was used; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 5.07, 95% CI 2-sided [2.47 to 10.40] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 9.46, 95% CI 2-sided [4.36 to 20.51] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 16.09, 95% CI 2-sided [6.69 to 38.73] — Survodutide 6.0 mg vs. Placebo
Statistical Analysis 4: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — Logistic regression estimates were used as input for the MCP-Mod. The logistic regression model was fitted without an intercept and included presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3] and the dose group as factors, and baseline liver fat content (assessed by MRI-PDFF) as a continuous linear covariate. P-values from the contrast tests corresponding to each dose response pattern evaluated were adjusted for the multiple comparisons performed; p < 0.0001, MCP-Mod linear model fit; Linear model fit assumption
Statistical Analysis 5: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p < 0.0001, MCP-Mod exponential-1 model fit; Model assumption: 25% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 6: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — Logistic regression estimates were used as input for the MCP-Mod. The logistic regression model was fitted without an intercept, and included presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3] and the dose group as factors, and baseline liver fat content (assessed by MRI-PDFF) as a continuous linear covariate. P-values from the contrast tests corresponding to each dose response pattern evaluated were adjusted for the multiple comparisons performed; p < 0.0001, MCP-Mod exponential-2 model fit; Model assumption: 5% of maximum effect achieved at dose 3.0 mg
Statistical Analysis 7: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p < 0.0001, MCP-Mod Emax1 model fit; Model assumption: 50% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 8: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 6]; p < 0.0001, MCP-Mod Emax2 model fit; Model assumption: 80% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 9: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Survodutide 4.8 mg - Actual Maintenance Treatment vs Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p < 0.0001, MCP-Mod quadratic model fit; Model assumption: Maximum effect is achieved at dose 4.8 mg

4. Secondary Outcome: Improvement of Liver Fat Content (Yes/ no) Defined as at Least 30% Relative Reduction in Liver Fat Content After 48 Weeks of Treatment Compared to Baseline Assessed by MRI-PDFF - Planned Maintenance Treatment
Description: Percentage of participants with improvement in liver fat content is reported. Improvement in liver fat content was defined as percentage reduction from baseline of ≥30% in liver fat content after 48 weeks of treatment compared to baseline.
  Liver fat content was assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF).
  Patients without post-baseline values were imputed as non-responders.
Time Frame: At baseline and at 48 weeks.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 73 | 72 | 74 | 74
Percentage of participants | 63.0 | 66.7 | 56.8 | 13.5
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; The logistic regression model included planned treatment, presence of diabetes of any type, baseline liver fat content and baseline fibrosis score. Firth's penalized regression was used; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 10.39, 95% CI 2-sided [4.60 to 23.45] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 4, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 12.06, 95% CI 2-sided [5.30 to 27.45] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 4, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 8.22, 95% CI 2-sided [3.66 to 18.50] — Survodutide 6.0 mg vs. Placebo
Statistical Analysis 4: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 6]; p < 0.0001, MCP-Mod linear model fit; Linear model fit assumption
Statistical Analysis 5: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p = 0.0031, MCP-Mod exponential-1 model fit; Model assumption: 25% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 6: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p = 0.0925, MCP-Mod exponential-2 model fit; Model assumption: 5% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 7: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p < 0.0001, MCP-Mod Emax1 model fit; Model assumption: 50% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 8: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 4]; p < 0.0001, MCP-Mod Emax2 model fit; Model assumption: 80% of maximum effect is achieved at dose 3.0 mg
Statistical Analysis 9: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Survodutide 4.8 mg - Planned Maintenance Treatment vs Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 3, analysis 6]; p < 0.0001, MCP-Mod quadratic model fit; Model assumption: Maximum effect is achieved at dose 4.8 mg

5. Secondary Outcome: Absolute Change of Liver Fat Content From Baseline After 48 Weeks of Treatment Assessed by MRI-PDFF - Actual Maintenance Treatment
Description: Absolute change of liver fat content (percentage [%]) from baseline after 48 weeks of treatment is reported. Liver fat content was assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF).
  Least Squares Mean (Standard error) were calculated from mixed-effect model for repeated measures (MMRM) including fixed effects for baseline liver fat content (%) as a continuous linear covariate, and treatment, presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3], visit, treatment by visit interaction and baseline by visit interaction as factors.
Time Frame: MMRM included measurements from baseline and at Week 28 and at Week 48 after first drug administration. MMRM estimates of absolute change from baseline to Week 48 is reported.
Population: Treated set - actual maintenance treatment. Patients are analyzed according to the actual treatment they received at the start of the dose maintenance period (for patients who reached the maintenance period) or the next maintenance dose up from the dose at treatment discontinuation (for patients who discontinued treatment prior to the maintenance period). The reported number of participants analyzed reflects the number of participants in the analysis model.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of liver fat content
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 68 | 60 | 51 | 73
percentage of liver fat content | -10.48 [-11.92 to -9.04] | -12.80 [-14.32 to -11.28] | -12.96 [-14.62 to -11.30] | -1.89 [-3.26 to -0.51]
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; Least Squares Mean differences and 95% confidence interval were calculated from mixed-effect model for repeated measures (MMRM) including fixed effects for baseline liver fat content (%) as a continuous linear covariate, and treatment, presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3], visit, treatment by visit interaction and baseline by visit interaction as factors; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -8.59, 95% CI 2-sided [-10.59 to -6.60] — "Survodutide 2.4 mg" - "Placebo"
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -10.91, 95% CI 2-sided [-12.96 to -8.86] — "Survodutide 4.8 mg" - "Placebo"
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -11.07, 95% CI 2-sided [-13.23 to -8.92] — "Survodutide 6.0 mg" - "Placebo"

6. Secondary Outcome: Absolute Change of Liver Fat Content From Baseline After 48 Weeks of Treatment Assessed by MRI-PDFF - Planned Maintenance Treatment
Description: Absolute change of liver fat content from baseline after 48 weeks of treatment is reported. Liver fat content was assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF).
  Least Squares Mean (Standard error) were calculated from mixed-effect model for repeated measures (MMRM) including fixed effects for baseline liver fat content (%) as a continuous linear covariate, and treatment, presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3], visit, treatment by visit interaction and baseline by visit interaction as factors.
Time Frame: as for outcome 5
Population: Treated set - planned maintenance treatment. Patients are analyzed for this endpoint according to the planned treatment (planned maintenance dose strength) they were assigned at randomisation even if patients did not reach the maintenance period at all, and therefore did not "settle" on any maintenance dose. The reported number of participants analyzed reflects the number of participants in the analysis model.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of liver fat content
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 61 | 64 | 58 | 69
percentage of liver fat content | -10.73 [-12.25 to -9.22] | -12.40 [-13.90 to -10.91] | -12.48 [-14.06 to -10.89] | -1.61 [-3.04 to -0.19]
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -9.12, 95% CI 2-sided [-11.21 to -7.03] — "Survodutide 2.4 mg" - "Placebo"
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -10.79, 95% CI 2-sided [-12.85 to -8.73] — "Survodutide 4.8 mg" - "Placebo"
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -10.86, 95% CI 2-sided [-13.00 to -8.73] — "Survodutide 6.0 mg" - "Placebo"

7. Secondary Outcome: Percent Change of Liver Fat Content From Baseline After 48 Weeks of Treatment Assessed by MRI-PDFF - Actual Maintenance Treatment
Description: Percent change of liver fat content (percentage [%]) from baseline after 48 weeks of treatment is reported. Liver fat content was assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF).
  Least Squares Mean (Standard error) were calculated from mixed-effect model for repeated measures (MMRM) including fixed effects for baseline liver fat content (%) as a continuous linear covariate, and treatment, presence of diabetes of any type [yes, no], baseline fibrosis score [F1, F2, F3], visit, treatment by visit interaction and baseline by visit interaction as factors.
Time Frame: MMRM included measurements from baseline and at Week 28 and at Week 48 after first drug administration. MMRM estimates of percent change from baseline to Week 48 is reported.
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change of liver fat content
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 68 | 60 | 51 | 73
percent change of liver fat content | -50.92 [-58.05 to -43.80] | -62.79 [-70.26 to -55.32] | -64.30 [-72.48 to -56.12] | -7.28 [-14.06 to -0.50]
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -43.64, 95% CI 2-sided [-53.49 to -33.79] — "Survodutide 2.4 mg" - "Placebo"
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -55.52, 95% CI 2-sided [-65.61 to -45.42] — "Survodutide 4.8 mg" - "Placebo"
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -57.02, 95% CI 2-sided [-67.66 to -46.39] — "Survodutide 6.0 mg"-"Placebo"

8. Secondary Outcome: Percent Change of Liver Fat Content From Baseline After 48 Weeks of Treatment Assessed by MRI-PDFF - Planned Maintenance Treatment
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Treated set - planned maintenance treatment: all patients that administered survodutide or placebo matching survodutide. Patients are analyzed for this endpoint according to the planned treatment (planned maintenance dose strength) they were assigned at randomisation even if patients did not reach the maintenance period at all, and therefore did not "settle" on any maintenance dose.
  The reported number of participants analyzed reflects the number of participants in the analysis model.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change of liver fat content
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 61 | 64 | 58 | 69
percent change of liver fat content | -52.20 [-59.66 to -44.75] | -60.82 [-68.16 to -53.48] | -61.97 [-69.78 to -54.16] | -5.71 [-12.70 to 1.28]
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -46.49, 95% CI 2-sided [-56.74 to -36.25] — "Survodutide 2.4 mg" - "Placebo"
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -55.11, 95% CI 2-sided [-65.25 to -44.98] — "Survodutide 4.8 mg" - "Placebo"
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 5, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p < .0001, MMRM — The p-value reported is considered nominal; Mean Difference (Net) = -56.26, 95% CI 2-sided [-66.76 to -45.77] — "Survodutide 6.0 mg"-"Placebo"

9. Secondary Outcome: Improvement of Fibrosis (Yes/ no) Defined as at Least One Stage Decrease in Fibrosis Stage After 48 Weeks of Treatment Assessed by Liver Biopsy - Actual Maintenance Treatment
Description: Percentage of participants with improvement of liver fibrosis is reported. Improvement of fibrosis was defined as at least one stage decrease in fibrosis stage after 48 weeks of treatment assessed by liver biopsy.
  The total score for the fibrosis stage ranges from 0 to 4 with higher score indication worsening of the disease and the stages of fibrosis based on their location are the following:
  * 1A Zone 3, perisinusoidal, delicate;
  * 1B Zone 3, perisinusoidal, dense;
  * 1C Portal, periportal only;
  * 2 Zone 3, perisinusoidal + portal, periportal only;
  * 3 Bridging fibrosis;
  * 4 Cirrhosis. For analysis purposes no distinction was made between stages 1A, 1B and 1C.
Time Frame: At baseline and after 48 weeks of treatment.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 93 | 69 | 52 | 79
Percentage of participants | 30.1 | 34.8 | 44.2 | 21.5
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.1894, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.79 to 3.26] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0685, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.95 to 4.20] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Actual Maintenance Treatment vs Placebo - Actual Maintenance Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0028, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.52 to 7.45] — Survodutide 6.0 mg vs. Placebo

10. Secondary Outcome: Improvement of Fibrosis (Yes/ no) Defined as at Least One Stage Decrease in Fibrosis Stage After 48 Weeks of Treatment Assessed by Liver Biopsy - Planned Maintenance Treatment
Description: as for outcome 9
Time Frame: At baseline and after 48 weeks of treatment.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 73 | 72 | 74 | 74
Percentage of participants | 34.2 | 36.1 | 33.8 | 21.6
Statistical Analysis 1: Comparison: Survodutide 2.4 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; The logistic regression model included planned treatment, presence of diabetes of any type and baseline fibrosis score. Firth's penalized regression was used; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0663, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.95 to 4.27] — Survodutide 2.4 mg vs. Placebo
Statistical Analysis 2: Comparison: Survodutide 4.8 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 10, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0672, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.95 to 4.23] — Survodutide 4.8 mg vs. Placebo
Statistical Analysis 3: Comparison: Survodutide 6.0 mg - Planned Maintenance Treatment vs Placebo - Planned Maintenance Treatment; [analysis description as in outcome 10, analysis 1]; Test type: Other — No confirmatory hypothesis testing was performed; p = 0.0512, Regression, Logistic — The p-value reported is considered nominal; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.00 to 4.46] — Survodutide 6.0 mg vs. Placebo

11. Secondary Outcome: Absolute Change From Baseline in NAS After 48 Weeks of Treatment Assessed by Liver Biopsy - Actual Maintenance Treatment
Description: Absolute change from baseline in NAS after 48 weeks of treatment assessed by liver biopsy is reported.
  The non-alcoholic fatty liver disease (NAFLD) activity score (NAS) represents the sum of subscores for steatosis (scored from 0-3), lobular inflammation (scored from 0-3) and ballooning (scored from 0-2), and the total score ranges from 0 to 8 with higher scores representing worsening of the disease.
Time Frame: At baseline and 48 weeks of treatment.
Population: Treated set - actual maintenance treatment. Patients are analyzed according to the actual treatment they received at the start of the dose maintenance period (for patients who reached the maintenance period) or the next maintenance dose up from the dose at treatment discontinuation (for patients who discontinued treatment prior to the maintenance period). Only patients with NAS data at baseline and at 48 weeks after treatment are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
Number analyzed (Participants) | 56 | 53 | 44 | 66
units on a scale | -2.8 (1.8) | -3.2 (1.8) | -3.3 (2.0) | -0.4 (1.6)

12. Secondary Outcome: Absolute Change From Baseline in NAS After 48 Weeks of Treatment Assessed by Liver Biopsy - Planned Maintenance Treatment
Description: as for outcome 11
Time Frame: At baseline and 48 weeks of treatment.
Population: Treated set - planned maintenance treatment: included all patients that were administered survodutide or placebo matching survodutide. Patients are analyzed for this endpoint according to the planned treatment (planned maintenance dose strength) they were assigned at randomisation even if patients did not reach the maintenance period at all, and therefore did not "settle" on any maintenance dose. Only patients with NAS data at baseline and at 48 weeks after treatment are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Survodutide 2.4 mg - Planned Maintenance Treatment | Survodutide 4.8 mg - Planned Maintenance Treatment | Survodutide 6.0 mg - Planned Maintenance Treatment | Placebo - Planned Maintenance Treatment
Number analyzed (Participants) | 53 | 55 | 48 | 63
units on a scale | -2.8 (1.8) | -3.2 (1.8) | -3.3 (1.9) | -0.2 (1.5)

ADVERSE EVENTS:
Time Frame: [All-Cause Mortality], [Serious Adverse Events], [Other Adverse Events]: From first study drug administration until last study drug administration plus 28 days of residual effect period (REP), up to 365 days.
Description: Treated set - actual maintenance treatment: included all patients that were administered survodutide or placebo matching survodutide. Patients are analyzed according to the actual treatment they received at the start of the dose maintenance phase (for patients who reached the maintenance period) or the next maintenance dose up from the dose at treatment discontinuation (for patients who discontinued treatment prior to the maintenance period).
Arm/Group | Survodutide 2.4 mg - Actual Maintenance Treatment | Survodutide 4.8 mg - Actual Maintenance Treatment | Survodutide 6.0 mg - Actual Maintenance Treatment | Placebo - Actual Maintenance Treatment
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/69 | 0/52 | 0/79
Serious Adverse Events (participants affected / at risk) | 5/93 | 7/69 | 5/52 | 5/79
Other Adverse Events (participants affected / at risk) | 85/93 | 60/69 | 49/52 | 68/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Survodutide 2.4 mg - Actual Maintenance Treatment (N=93) | Survodutide 4.8 mg - Actual Maintenance Treatment (N=69) | Survodutide 6.0 mg - Actual Maintenance Treatment (N=52) | Placebo - Actual Maintenance Treatment (N=79)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Blindness transient (Eye disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Survodutide 2.4 mg - Actual Maintenance Treatment (N=93) | Survodutide 4.8 mg - Actual Maintenance Treatment (N=69) | Survodutide 6.0 mg - Actual Maintenance Treatment (N=52) | Placebo - Actual Maintenance Treatment (N=79)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 15 | 10 | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 12 | 5 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 16 | 12 | 15 | 14
Diarrhoea (Gastrointestinal disorders) | 38 | 37 | 29 | 20
Dyspepsia (Gastrointestinal disorders) | 14 | 6 | 11 | 3
Eructation (Gastrointestinal disorders) | 12 | 9 | 8 | 2
Flatulence (Gastrointestinal disorders) | 8 | 6 | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 7 | 3 | 5
Nausea (Gastrointestinal disorders) | 60 | 46 | 33 | 22
Vomiting (Gastrointestinal disorders) | 38 | 33 | 15 | 6
Asthenia (General disorders) | 5 | 1 | 2 | 1
Early satiety (General disorders) | 2 | 2 | 6 | 1
Fatigue (General disorders) | 18 | 10 | 8 | 7
Injection site bruising (General disorders) | 3 | 1 | 1 | 6
Injection site pain (General disorders) | 3 | 0 | 0 | 6
Injection site reaction (General disorders) | 3 | 3 | 1 | 5
Malaise (General disorders) | 2 | 1 | 5 | 0
Pyrexia (General disorders) | 4 | 3 | 2 | 5
COVID-19 (Infections and infestations) | 19 | 15 | 5 | 16
Influenza (Infections and infestations) | 2 | 2 | 2 | 5
Nasopharyngitis (Infections and infestations) | 6 | 12 | 4 | 10
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 2 | 3
Urinary tract infection (Infections and infestations) | 7 | 1 | 7 | 5
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 5
Lipase increased (Investigations) | 5 | 4 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 20 | 9 | 8 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 5
Dizziness (Nervous system disorders) | 11 | 5 | 3 | 6
Headache (Nervous system disorders) | 21 | 12 | 6 | 13
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT04771273/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT04771273/SAP_001.pdf